CLINICAL TRIAL: NCT02959372
Title: Lung Ultrasoung Guided Treatment in Chronic Heart Failure Patients: a Randomized Controlled Trial
Acronym: LUS-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IIBSP-ECO-2016-55
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- lung ultrasound group (Experimental): lung ultrasound results
  Interventions: Other: lung ultrasound
- control group (Placebo Comparator): The attending physician will not have the result of the lung ultrasound
  Interventions: Other: placebo

INTERVENTIONS:
Other: lung ultrasound
  Arms: lung ultrasound group
Other: placebo — lung ultrasound. The attending physician will not know the result
  Arms: control group

SUMMARY:
Introduction: Despite the great advances in treatment, heart failure (HF) continues to be an important health problem because of its high prevalence, morbidity, mortality and associated costs. Research shows at least 40% of HF in-patients are going to be readmitted in the following year. Thus, new strategies to reduce HF decompensations are needed.

In recent studies, pulmonary congestion which is expressed in the form of B-lines detected by lung ultrasound (LUS) has proven to be a potent prognostic predictor of hospitalization and mortality in HF. Moreover, the use of LUS is becoming more common due to its availability (with pocket devices with sizes approaching those of smart phones); its simplicity (rapid learning curve and rapid examination, less than 5 minutes) and its safety (radiation free).

We hypothesize that a management guided by LUS in HF patients may improve outcomes.

Objective: The aim of our study is to evaluate if ambulatory LUS guided treatment of patients after a hospitalization for HF, decreases the combined end-point of mortality or re-hospitalization after a 6 months follow-up.

Study design: The design of our study is a randomized, simple blinded, clinical trial.

Eligible patients are patients older than 18 years of age who have been hospitalized for HF. The exclusion criteria are life expectancy of less than 6 months or uninterpretable lung ultrasound. Eligible patients are going to be randomized into either the "LUS group" or the "control group".

The follow-up consists of visits to the HF clinic at periods of 15 days, 1, 3 and 6 months after the initial hospitalization. LUS is going to be performed on all patients despite their respective group. Only in relation to the "LUS group", the treating physician will have the result of the examination and the subsequent treatment adjustment could be made in response to those findings.

This study complies with the Declaration of Helsinki and the study protocol is being evaluated by the Ethic Committee of our institution.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Current hospitalization for heart failure decompensation

Exclusion Criteria:

* Not able to do the follow up
* Life expectancy of less than 6 months
* uninterpretable lung ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-11; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
mortality or re-hospitalization | 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eulalia Roig, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain